CLINICAL TRIAL: NCT02504463
Title: A Single-Center, Open-Label Study to Evaluate the Absorption, Metabolism, and Excretion of Single Doses of [14c]-Samidorphan in Healthy Male Subjects
Brief Title: A Study of [14c]-Samidorphan (Also Known as ALKS 33) in Healthy, Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK33-B107
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Alkermes; Samidorphan; ALKS 33; Healthy Volunteer; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Samidorphan IV (Experimental): Samidorphan solution for IV administration
  Interventions: Drug: Samidorphan IV
- Samidorphan sublingual (Experimental): [14c]-Samidorphan for sublingual administration
  Interventions: Drug: [14c]-Samidorphan sublingual
- Samidorphan oral (Experimental): [14c]-Samidorphan for oral administration
  Interventions: Drug: [14c]-Samidorphan oral

INTERVENTIONS:
Drug: Samidorphan IV — Single IV administration
  Arms: Samidorphan IV
Drug: [14c]-Samidorphan sublingual — Single sublingual administration containing radiolabel
  Arms: Samidorphan sublingual
Drug: [14c]-Samidorphan oral — Single oral administration containing radiolabel
  Arms: Samidorphan oral

SUMMARY:
This study will determine the pharmacokinetics (PK) of [14c]-samidorphan in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of greater than/equal to 19 and less than/equal to 32 kg/m^2 at screening (minimum weight of 50.0 kg)
* Generally good health
* Subjects must agree to reduce the risk of a female partner becoming pregnant during the study and for 30 days after the last dose of the study drug by abstinence from heterosexual relationships or use of a reliable contraceptive method
* Additional criteria may apply

Exclusion Criteria:

* Clinically significant illness within 30 days
* History of alcohol or opioid dependence, or positive urine toxicological screen for marijuana, cocaine, amphetamines, opioids, barbiturates, and benzodiazepines
* History of oral or gastrointestinal disease
* Irregular bowel or bladder function
* History of allergy or hypersensitivity to opioid medications or opioid antagonists (eg, naltrexone, naloxone)
* Current or pending legal charges or probation that would interfere with study conduct
* Use of alcohol within 24 hours prior to admission or urine positive test for alcohol at screening or admission
* Tobacco or nicotine use within 90 days
* Anticipated need for prescription medicines during the study period
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | Up to 120 hours after each dose
  Area under the concentration time curve of total radioactivity from time 0 to last observed concentration in blood and plasma
Cmax | Up to 120 hours after each dose
  Maximum concentration of total radioactivity in blood and plasma
Tmax | Up to 120 hours after each dose
  Time to maximum concentration of total radioactivity in blood and plasma
Fe%0-t | Up to 120 hours after each dose
  Fraction of dose excreted in urine and feces

SECONDARY OUTCOMES:
Safety and tolerability will be measured by the incidence of Adverse Events | Up to 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Stanford, MD, Study Director — Alkermes Medical Director
Locations (1):
- Alkermes Investigational Site, Austin, Texas, United States